CLINICAL TRIAL: NCT04098042
Title: Retrospective, Observational Register to Investigate the Procedural and Post Procedural Implantation of Bioabsorbable Magnesium Scaffolds MAGMARIS (MAGIC Registry)
Brief Title: MAGnesIum Alloy Scaffold for Coronary Artery Disease (MAGIC)
Acronym: MAGIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Collaborators: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, MD, San Luigi Gonzaga Hospital
Other Study IDs: 001/2019
Record Dates: First submitted 2019-09-09; First posted 2019-09-20 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: Bioresorbable scaffolds; Magnesium made bioresorbable scaffolds; Magmaris; coronary artery disease; Percutaneous coronary intervention; Myocardia infarction; multivessel coronary disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Scaffold: Patients receiving during PCI the implantation of at least one Magnesium Made Bioresorbable Scaffold "Magmaris"
  Interventions: Device: Scaffold

INTERVENTIONS:
Device: Scaffold — implantation of a Magmaris scaffold

SUMMARY:
The retrospective study will investigate the clinical performance and long-term safety of scaffold implantation in a real world setting including high volume PCI centers in Italy

DETAILED DESCRIPTION:
Coronary stents are the default devices for the treatment of coronary artery disease in percutaneous coronary intervention (PCI) according to existing guidelines. However, thrombosis and restenosis are still the main limitations of current permanent metallic stents. In contrast to Bare Metal Stents (BMSs), Drug Eluting Stents (DESs) have a reduced restenosis rate due to the presence of antiproliferative agents in the coating layer of the stent surface and reduced rate of repeat revascularisation. However, late and very late stent thrombosis remains the limitation of DES in spite of prolonged dual antiplatelet therapy. Bioabsorbable scaffolds have been introduced to overcome limitations of permanent metallic stents.

The aim of this observational retrospective study is to investigate the clinical performance and long-term safety of scaffold in a real world setting.

Institution involved in the present registry are high volume PCI centers. Operators have experience in PCI with bioresorbable scaffolds technology

The study organization is based on:

DATA SAFETY MONITORING BOARD (DSMB) All adverse events will be reported to the DSMB and reviewed on an on-going basis throughout the subject enrolment and follow-up period to ensure the safety of subjects enrolled in this study. In case of clinical events, coronary artery angiographies and percutaneous coronary interventions was reviewed by an independent core-lab.

ELIGIBILITY:
Inclusion Criteria:

* subjects >18 years
* Able to provide an informed consent
* implantation of at least one scaffold

Exclusion Criteria:

* inability to provide at least one year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease needing the treatment of de novo native coronary artery lesions.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2016-07-30 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Device Oriented Cardiac Events (DOCE) rate | 1 year
  Rate of DOCE, a composite of cardiovascular death, target vessel myocardial infarction and target lesion revascularization.

SECONDARY OUTCOMES:
Cardiac death rate | 1 year
  Rate of unexpected death due to cardiac causes
Target vessel myocardial infarction rate | 1 year
  Rate of myocardial infarction due to scaffold failure
Target lesion revascularization rate | 1 year
  rate of any revascularization of the lesion treated with a scaffold

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University Hospital of Ferrara, Cona, Ferrara
  - Interventional Unit, San Luigi Gonzaga University Hospital, Orbassano, and Rivoli Hospital, Turin, Italy, Turin

IPD SHARING:
Plan to Share IPD: Undecided